CLINICAL TRIAL: NCT03216096
Title: A Prospective, Open Label, One-arm, 4-weeks Study Assessing Safety and Efficacy of DE-089 Ophthalmic Solution in Patients With Dry Eye Disease -Phase 1 Study in Dry Eye Patients
Brief Title: Assessing Safety and Efficacy of DE-089 Ophthalmic Solution in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00891601
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3% DE-089 ophthalmic solution (Experimental)
  Interventions: Drug: Placebo ophthalmic solution and 3% DE-089 ophthalmic solution

INTERVENTIONS:
Drug: Placebo ophthalmic solution and 3% DE-089 ophthalmic solution — Placebo ophthalmic solution; 1 drop, 6 times daily (every 2-3 hours) instilled into both eyes for 2-week run-in period 3% DE-089 ophthalmic solution; ; 1 drop, 6 times daily (every 2-3 hours) instilled into both eyes for 4-week treatment period

SUMMARY:
The objective of this study is to assess safety and efficacy of DE-089 ophthalmic solution in patients with dry eye disease in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* At least 6-month dry eye history

Exclusion Criteria:

* Diagnosed with Stevens-Johnson Syndrome or ocular pemphigoid
* Diagnosed with keratoconjunctival chemical burns or thermal burn
* Eye disease other than dry eye disease which needs treatment
* Allergic conjunctivitis that may possibly be aggravated during the clinical study and inappropriate for efficacy evaluation
* Those who need to wear contact lenses during the clinical study
* Those who are considered inappropriate for this study by the investigator or subinvestigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining score | Week 4
  Change in corneal fluorescein staining score at week 4/ at the time of discontinuation

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Keelung Chang Gung Memorial Hospital, Keelung
  - National Taiwan University Hospital, Taipei